CLINICAL TRIAL: NCT00826384
Title: Phase 1,Single-blind, Randomized, Controlled Study to Evaluate the Safety and Effectivity of TACE Therapy of HCC(Hepatocellular Carcinoma) With Blocking Tumor Blood Temporarily and Enhancing Perfu
Brief Title: Transarterial Chemoembolization (TACE) Therapy of Hepatocellular Carcinoma (HCC) With Blocking Tumor Blood Temporarily and Enhancing Perfusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-001
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; transcatheter arterial chemoembolization; overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: balloon catheter — transcatheter arterial chemoembolization therapy with balloon catheter

SUMMARY:
According to radiology imaging, the patients of HCC are divided into two groups(hypovascular tumor group and moderately vascular tumor group). Every group is divided into TACE therapy with balloon catheter subgroup and regular TACE therapy subgroup. Patients take the TACE therapy each 45 days, and have MRI diffusion examine or CT one week before next therapy. All objects are observed until the end event happening or in the group for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* sign the written informed consent form provided.
* diagnosed clinically as HCC,need to take TACE.

Exclusion Criteria:

* have had an allergic reaction following iodine.
* have been in any TACE or radiotherapy or biotherapy within 30 days before the study.
* HCC of diffuse type,failure of hepatic function, chronic illness or disease including failure of heart function, uncontrolled high blood pressure, heart disorders, serious infection, uncontrolled diabetes mellitus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD, Study Chair — Eastern hepatobilliary surgery hospital
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China